CLINICAL TRIAL: NCT03976791
Title: A Randomized Controlled Study of Phacoemulsification by the Enlarged Internal Incision and the Regular 2.2mm Incision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019KYPJ078
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enlarged internal incision (Experimental): enlarged the internal incision about 0.4mm
  Interventions: Procedure: enlarged internal incision
- Regular 2.2mm incision (Placebo Comparator): regular 2.2mm corneal incision for microincision coaxial phacoemulsification
  Interventions: Procedure: regular 2.2mm incision

INTERVENTIONS:
Procedure: enlarged internal incision — enlarging the internal incision about 0.4mm
  Arms: Enlarged internal incision
Procedure: regular 2.2mm incision — 2.2mm microincision coaxial phacoemulsification
  Arms: Regular 2.2mm incision

SUMMARY:
Objective and Principle: To evaluate whether enlarging the incision can reduce corneal complications associated with phacoemulsification with regular 2.2 mm incision.

The aim of this study: To evaluate whether the technique of enlarging internal incision could reduce the incidence of descemet membrane detachment after 2.2 mm incision phacoemulsification.

Secondary outcome: To evaluate whether the technique of enlarged internal incision can reduce other corneal complications such as corneal edema and astigmatism after 2.2 mm incision phacoemulsification.

Study Design: A prospective randomized controlled study

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract patients
* Age from 65 to 90
* The diameter of pupil after mydriasis is more than 6 mm
* LOCS III nuclear grade ≥4
* Corneal endothelial cell count > 1500 cells/mm2
* Phacoemulsification and intraocular lens implantation are planned
* Agree to participate in this study and sign informed consent

Exclusion Criteria:

* History of ocular trauma
* Anterior segment lesions (exfoliation syndrome, suspension ligament injury or relaxation, corneal and iris lesions, glaucoma)
* Other ocular diseases that impair visual function, such as optic neuropathy, uveitis and ocular tumors
* History of Ophthalmic Surgery
* Intraoperative and Postoperative Complications

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
descemet membrane detachment(DMD) | postoperative 1 week
  DMD at the incision observed by anterior segment optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Doctor, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China